CLINICAL TRIAL: NCT06304155
Title: Application of FDG Combined With FAPI PET Dual Imaging in the Diagnosis and Staging of Oropharyngeal and Laryngeal Cancer
Status: Recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 202437
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic efficacy,SUV — The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 18F-FAPI PET were calculated and compared to evaluate the diagnostic efficacy.
  Standardized uptake value (SUV) of 18F-FDG and 18F-FAPI for each target lesion of subject or suspected primary tumor or/and metastasis.

SUMMARY:
According to statistics, in 2020, new head and neck malignancies in the world accounted for 4.9% (931931 cases) of malignant tumors in the whole body, and the new death cases were 467125, accounting for 4.7% of malignant tumors in the whole body. The high incidence rate and mortality brought great burden to the medical system. In addition, due to various types of head and neck cancer, hidden location, impact on function and quality of life, and low overall survival rate, this type of disease has seriously threatened human health and social development. The incidence of oropharyngeal cancer and laryngeal cancer is more subtle. Traditional examination methods include CT(computer tomography), MR(magnetic resonance), and laryngoscopy, but they cannot make accurate judgments on the systemic TNM(primary tumor, regional nodes, metastasis) staging of oropharyngeal cancer and laryngeal cancer. 18F-FDG(18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET/CT examination can better diagnose and stage compared to traditional examination methods. However, due to the interference of more inflammatory lesions or physiological uptake in the pharynx, the false positive rate of 18F-FDG PET/CT examination is significantly increased, 18F-FAPI(18F-fibroblast activation protein inhibitors) is a novel broad-spectrum tumor imaging agent that can be specifically uptake by fibroblasts in the tumor microenvironment, and has lower physiological uptake and acute inflammatory lesion uptake in the larynx. 18F-FAPI PET/CT examination can more accurately stage tumors throughout the body than 18F-FDG PET/CT examination. Combined with PET/MR local scanning, it will further improve the accuracy of T and N staging of local tumors. Therefore, It is of great significance for clinical diagnosis and treatment to effectively and reliably determine the systemic TNM staging of oropharyngeal and laryngeal cancer through non-invasive methods.

DETAILED DESCRIPTION:
This study is a prospective, single study and has been approved by the ethics committee. The subjects of this studywere from January 1,2024 to January 1,2026.The detailed description is as follows:

1. Patients: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "Eligibility Criteria" column.
2. Clinical data collection: Record the course of disease, CT examination, MR examination, laryngoscopy examination, PET/CT examination, PET/MR examination, and other information of all patients.
3. CT or MRI image analysis: Record the location and number of lesions, measure the long diameter of the primary and metastatic lesions, and the short diameter of lymph nodes on CT or MRI images.
4. PET image analysis: Record and evaluate the following indicators:

   the maximum, mean and peak standardized uptakevalue (SUVmax, SUVmean and SUVpeak), Metabolic lesion volume (MLV), total lesion glycolysis (TLG).
5. Statistical analysis: Use descriptive statistical methods to compare the age of patients and the standardized uptake values of FDG and FAPI. Normal distribution data is represented as mean ± standard deviation, while non normal distribution data is represented as median with IQR. Compare the normal distribution data between two groups using paired two sample t-test, and compare the non normal distribution data between two groups using McNemar test. Using a four grid table McNemar χ Compare the diagnostic efficacy of 18F-FDG PET and 18F-FAPI PET through 2 tests, calculate and compare the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of 18F-FDG and 18F-FAPI PET. Due to the potential impact of tumor type on diagnosis, subgroup analysis was conducted on the diagnostic efficacy of 18F-FDG PET and 18F-FAPI PET. Due to the possibility of multiple metastatic lesions in a given participant, the diagnostic results may be correlated within the participant. Therefore, sensitivity analysis of metastatic lesions is also performed based on a generalized linear mixed effects model by combining this correlation between different lesions within the same participant. Double tailed P<0.05 indicates a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high clinical suspicion of oropharyngeal and laryngeal cancer: CT and MR examinations reveal space occupying lesions in the oropharynx and laryngopharynx, with high suspicion of laryngeal cancer;
2. Recently diagnosed patients: patients who have recently been diagnosed with oropharyngeal cancer and laryngeal cancer, have not undergone surgical resection but are willing to undergo surgery;
3. Patients who have been diagnosed with oropharyngeal and laryngeal cancer and have undergone concurrent radiotherapy, chemotherapy, or immunotherapy, and are preparing to undergo preoperative staging in the near future;
4. Patients with high suspicion of oropharyngeal and laryngeal cancer through imaging examination, and later confirmed by pathology as non oropharyngeal or laryngeal cancer;
5. Patient age ≥ 18 years old;
6. The patient voluntarily participates and signs an informed consent form.

Exclusion Criteria:

1. Patients who refuse to undergo surgery;
2. Patients highly suspected of lymphoma or metastasis in clinical or imaging studies;
3. Patients with multiple neck metastases identified through imaging examination that cannot be surgically treated;
4. Patients with malignant tumors in other parts of the body found through imaging examination that cannot be operated on;
5. Pregnancy or lactation period;
6. The imaging quality is poor and cannot be used for diagnosis and evaluation;
7. Patients with contraindications for MR examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "EligibilityCriteria" colymn.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | Completed within half year after end of the study
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 18F-FAPI PET were calculated and compared to evaluate the diagnostic efficacy.

SECONDARY OUTCOMES:
SUV | Completed within half year after end of the study
  Standardized uptake value (SUV) of 18F-FDG and 18F-FAPI for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steuer CE, El-Deiry M, Parks JR, Higgins KA, Saba NF. An update on larynx cancer. CA Cancer J Clin. 2017 Jan;67(1):31-50. doi: 10.3322/caac.21386. Epub 2016 Nov 29. PMID 27898173
- [Derived] Xia R, Wang X, Cheng J, Li X, Sun J, Zeng Q, Hu D, You J, Xiong Y, Chen X. Head-to-head comparison of [18F]FAPI-42 and [18F]FDG PET/CT in the evaluation of laryngeal squamous cell carcinoma. Eur J Nucl Med Mol Imaging. 2025 Jul;52(9):3101-3113. doi: 10.1007/s00259-025-07180-8. Epub 2025 Mar 8. PMID 40055207
- See also: An Update on Larynx Cancer — http://pubmed.ncbi.nlm.nih.gov/27898173/